CLINICAL TRIAL: NCT00562965
Title: An Open-label, Randomized, Phase 3 Study Of Inotuzumab Ozogamicin (Cmc-544) Administered In Combination With Rituximab Compared To A Defined Investigator's Choice Therapy In Subjects With Relapsed Or Refractory, Cd22- Positive, Follicular B-cell Non Hodgkin's Lymphoma
Brief Title: Study Comparing Inotuzumab Ozogamicin In Combination With Rituximab Versus Defined Investigator's Choice In Follicular Non-Hodgkin's Lymphoma (NHL)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 3129K4-3301; B1931006 (Other: Alias Study Number); 2007-000219-27 (EudraCT Number)
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Results first posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-12

CONDITIONS: Lymphoma, Follicular
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Inotuzumab Ozogamicin; Rituximab; Cyclophosphamide; Vincristine; Prednisone; Prednisolone; Mitoxantrone; fludarabine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Subjects will receive rituximab intravenously at a dose level of 375 mg/m² on day 1 of each cycle followed by inotuzumab ozogamicin administered intravenously at a dose level of 1.8 mg/m2 on day 2. The sequence will be repeated every 28 days.
  Interventions: Drug: inotuzumab ozogamicin; Drug: rituximab
- B (Active Comparator): Subjects will receive the investigator's choice from the following rituximab-containing regimens: R-CVP or R-FND. The investigator's choice of therapy will be administered every 21 days. Dosing for R-CVP will be intravenous rituximab at a dose of 375 mg/m2 on day 1, intravenous cyclophosphamide at a dose of 750 mg/m2 on day 1, intravenous vincristine at a dose of 1.4 mg/m2 (not to exceed 2 mg) on day 1, and oral prednisone/prednisolone at a dose of 40 mg/m2 on days 1 through 5. Dosing for R-FND will be as follows: rituximab 375 mg/m2 intravenous on day 1, mitoxantrone 10 mg/m2 intravenous on day 2, fludarabine 25 mg/m2 intravenous on days 2 through 4 and oral dexamethasone 20 mg/day on days 1-5.
  Interventions: Drug: rituximab; Drug: cyclophosphamide; Drug: vincristine; Drug: prednisone/prednisolone; Drug: mitoxantrone; Drug: fludarabine; Drug: dexamethasone

INTERVENTIONS:
Drug: inotuzumab ozogamicin — IV administration, 1.8mg/m² on day 2 of each cycle every 28 days, for up to 8 cycles.
  Arms: A
Drug: rituximab — IV administration, 375 mg/m² on day 1 of each cycle every 28 days, for up to 8 cycles.
  Arms: A
Drug: rituximab — intravenous rituximab at a dose of 375 mg/m2 on day 1
  Arms: B
Drug: cyclophosphamide — intravenous cyclophosphamide at a dose of 750 mg/m2 on day 1
  Arms: B
Drug: vincristine — intravenous vincristine at a dose of 1.4 mg/m2 (not to exceed 2 mg) on day 1
  Arms: B
Drug: prednisone/prednisolone — oral prednisone/prednisolone at a dose of 40 mg/m2 on days 1 through 5
  Arms: B
Drug: mitoxantrone — mitoxantrone 10 mg/m2 intravenous on day 2
  Arms: B
Drug: fludarabine — fludarabine 25 mg/m2 intravenous on days 2 through 4
  Arms: B
Drug: dexamethasone — oral dexamethasone 20 mg/day on days 1-5
  Arms: B

SUMMARY:
This protocol is designed to assess the efficacy and safety of inotuzumab ozogamicin given with rituximab compared to a defined investigator's choice therapy. Subjects will be randomized to one of these two arms of the study.

DETAILED DESCRIPTION:
On January 14th 2009, enrollment in the study was discontinued because of poor enrollment and because it was unlikely that the study would meet the estimated enrollment of approximately 978 subjects. The decision was not prompted by the identification of any safety signals in this or other studies. Active treatment and follow-up of the already enrolled subjects was continued. On July, 22th 2010 , the study was amended to shorten the long-term follow-up to one year after active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of CD20 and CD22-positive, follicular lymphoma, who have received 1 or 2 prior regimens, at least 1 of which should have contained administration of rituximab (either as a single agent or in combination).
* Age 18 years or older.
* ECOG performance status <= 2.
* ANC >= 1.5 x 10^9/L (1500/mL) and platelets >= 75 x 10^9/L (75,000/mL), serum creatinine <= 1.5 x ULN and urine protein to creatinine ratio of <= 0.5, total bilirubin <= 1.5 x ULN, AST and ALT <= 2.5 x ULN.
* At least 1 measurable disease lesion that is >= 1.5 cm x 1.5 cm by CT or MRI, in an area of no prior radiation therapy, or documented progression in an area that was previously irradiated.

Exclusion Criteria:

* Subjects with clinical evidence of transformation to a more aggressive subtype of lymphoma or grade 3b follicular lymphoma.
* Subjects whose disease is rituximab refractory, meaning that they did not have a CR or PR, or that they experienced disease progression within 6 months from the initiation of the rituximab or rituximab containing treatment regimen administered immediately preceding study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (39):
- United States (17):
  - Facey Medical Group, Mission Hills, California
  - Deaconess Clinic, Evansville, Indiana
  - The Harry & Jeanette Weinberg Cancer Inst at Franklin Square, Baltimore, Maryland
  - Newland Medical Associates, Novi, Michigan
  - Newland Medical Associates, PC, Southfield, Michigan
  - Park Nicollet Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Hematology and Oncology Associates, Columbus, Mississippi
  - Hematology and Oncology Associates, Corinth, Mississippi
  - Hematology and Oncology Associates at Bridgepoint, Tupelo, Mississippi
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Hematology Oncology Associates of Northern New Jersy, Morristown, New Jersey
  - Advanced Oncology Associates, Armonk, New York
  - Advanced Oncology Associates, New Rochelle, New York
  - Marc Zimmerman, MD, Pomona, New York
  - Avi Einzing, MD, The Bronx, New York
  - Wenatchee Valley Medical Center, Wenatchee, Washington
- Centro de Transplantes de medula Osea de Rosario, CETRAMOR, Rosario, Santa Fe Province, Argentina
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - Oncologisch Centrum GZA - Location St. Augustinus, Wilrijk
- Canada (4):
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - C.H.A. Enfant-Jesus, Québec, Quebec
  - CHUS-Hopital Fleurimont, Sherbrooke, Quebec
- Hong Kong (2):
  - Prince of Wales Hospital, Shatin, NEW Territories
  - Queen Mary Hospital, Hong Kong
- India (3):
  - Jehangir Clinical Development Centre, Pune, Maharashtra
  - MMF Joshi Hospital and Ratna Memorial Hospital, Pune, Maharashtra
  - B. P. Poddar Hospital and Medical Research Ltd., Kolkata, West Bengal
- Divisione di Ematologia - Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
- Hospital Universitario de Nuevo Leon, Monterrey, Nuevo León, Mexico
- Instytut Hematologii i Transfuzjologii, Warsaw, Poland
- Hospitais Da Universidade De Coimbra, Coimbra, Portugal
- Moscow Regional Research Clinical Institute named after Vladimirsky, Moscow, Russia
- Wits Donald Gordon Clinical Trial Site, Johannesburg, Gauteng, South Africa
- Yonsei University Health System-Severance Hospital, Seoul, South Korea
- Spain (3):
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Santa Creu I Sant Pau, Barcelona
  - Hospital de La Princesa, Madrid

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3129K4-3301&StudyName=Study%20Comparing%20Inotuzumab%20Ozogamicin%20In%20Combination%20With%20Rituximab%20Versus%20Defined%20Investigator%27s%20Choice%20In%20Follicular%20Non-Hodgkin%27s%20Lymp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of participants started on 15 November 2007 and completed on 16 January 2009. The trial was terminated (07 April 2011) due to poor accrual of 29 out of 978 planned participants.
Groups:
- Rituximab + Inotuzumab Ozogamicin: Participants received intravenous infusion of rituximab 375 milligram per square meter (mg/m^2) of body surface area (BSA) on Day 1 followed by intravenous infusion of inotuzumab ozogamicin (CMC-544) 1.8 mg/m^2 of BSA on Day 2 for each cycle up to 8 cycles. Each cycle was of 28 days.
- Control Regimens R-CVP + R-FND: Participants received either regimen containing intravenous infusion of rituximab 375 mg/m^2 of BSA along with intravenous infusion of cyclophosphamide 750 mg/m^2 of BSA and vincristine 1.4 mg/m^2 of BSA on Day 1 followed by oral prednisone/prednisolone 40 mg/m^2 of BSA on Days 1 through 5 for up to 8 cycles (R-CVP); or regimen containing intravenous infusion of rituximab 375 mg/m^2 of BSA on Day 1 followed by intravenous infusion of novantrone (mitoxantrone) 10 mg/m^2 of BSA on Day 2, intravenous infusion of fludarabine 25 mg/m^2 of BSA on Days 2 through 4, and oral dexamethasone 20 mg once daily on Days 1 through 5 for up to 8 cycles (R-FND). Each regimen cycle was of 21 days.
Period: Overall Study
Arm/Group | Rituximab + Inotuzumab Ozogamicin | Control Regimens R-CVP + R-FND
Started | 15 | 14
Treated | 15 | 13
Completed | 12 | 8
Not Completed | 3 | 6
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 2 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population included all participants who were randomized in to the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab + Inotuzumab Ozogamicin | Control Regimens R-CVP + R-FND | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (11.4) | 60.9 (12.4) | 61.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from randomization to disease progression or death due to any cause, whichever occurred first, censored at the last tumor evaluation date. PFS calculated as (Months) = (first event date minus randomization date plus 1) divided by 30.44.
Time Frame: Baseline until disease progression or death or up to 1 year after last dose of study drug
Population: Intent-to-treat population included all participants who were randomized in to the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Inotuzumab Ozogamicin | Control Regimens R-CVP + R-FND
Number analyzed (Participants) | 15 | 14
months | NA [22.2 to NA] — Median and upper limit of confidence interval was not estimable because majority of participants were censored. | 16.4 [7.9 to 28.4]
Statistical Analysis 1: Comparison: Rituximab + Inotuzumab Ozogamicin vs Control Regimens R-CVP + R-FND; To detect a hazard ratio of 0.77 with 85% power using a 2-sided log-rank test at the 5% significance level, it was planned that approximately 978 participants were needed to be randomized but due to premature termination only 29 participants were randomized; Test type: Superiority or Other; p = 0.0358, Cox proportional hazard regression model; A 2-sided 5% significance level on a stratified Cox proportional hazard regression model was used; Hazard Ratio (HR) = 0.19, 95% CI 2-sided [0.04 to 1.02] — In this regression model, treatment arm was the covariate and the strata (number of prior regimens, investigator's choice of therapy and geographical region) over which participants were stratified prior to randomization were the variables

2. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: OR was based on assessment of complete response(CR),unconfirmed CR(Cru),partial response(PR) as per International Response Criteria for Non-Hodgkin's Lymphoma.Confirmed response=response persists on repeat imaging at least 4 weeks after initial response.CR=complete disappearance of all detectable clinical/radiographic evidence of disease,lymph nodes regressed to normal size [at least 1.5 centimeter(cm) or less],spleen regressed,not palpable on physical examination,bone marrow infiltrate cleared on repeat aspiration/biopsy.PR=at least 50 percent (%) decrease in sum of product diameters of 6 greatest dominant nodes,no increase in other nodes,liver/spleen,no new sites of disease. CRu=residual lymph node greater than 1.5 cm in transverse diameter that has regressed more than 75% in product diameter.Individual nodes previously confluent,regressed more than 75% in product diameters.Indeterminate bone marrow (increased number/size of lymph aggregates without cytologic/architectural atypia).
Time Frame: Baseline, every 6 to 12 weeks during treatment period, end of treatment (EOT) (42 days after last dose), every 12 weeks during follow-up for up to 1 year after the last dose of study drug
Population: Intent-to-treat population included all participants who were randomized in to the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab + Inotuzumab Ozogamicin | Control Regimens R-CVP + R-FND
Number analyzed (Participants) | 15 | 14
percentage of participants | 93.3 [68.1 to 99.8] | 64.3 [35.1 to 87.2]
Statistical Analysis 1: Comparison: Rituximab + Inotuzumab Ozogamicin vs Control Regimens R-CVP + R-FND; Test type: Superiority or Other; p = 0.0801, Fisher Exact

3. Secondary Outcome: Overall Survival Probability at Months 6, 12 and 24
Description: Overall survival was defined as the time from randomization to death due to any cause, censoring at the date of last contact or the end of the study. Participants who withdrew or lost to follow-up from study without having death documented were censored at the date of last contact. Kaplan-Meier estimates of the probability of survival at 6, 12 and 24 months was used to estimate the survival function.
Time Frame: Baseline up to Month 6, 12, 24
Population: Intent-to-treat population included all participants who were randomized in to the study.
Measure: Number (95% Confidence Interval); unit: percent chance of survival
Arm/Group | Rituximab + Inotuzumab Ozogamicin | Control Regimens R-CVP + R-FND
Number analyzed (Participants) | 15 | 14
percent chance of survival
  Overall Survival: Baseline up to Month 6 | 100.0 [100.0 to 100.0] | 92.3 [77.8 to 100.0]
  Overall Survival: Baseline up to Month 12 | 86.7 [69.5 to 100.0] | 83.9 [63.4 to 100.0]
  Overall Survival: Baseline up to Month 24 | 86.7 [69.5 to 100.0] | 67.1 [40.7 to 93.6]
Statistical Analysis 1: Comparison: Rituximab + Inotuzumab Ozogamicin vs Control Regimens R-CVP + R-FND; Test type: Superiority or Other; p = 0.1727, Cox proportional hazard regression model; Stratified Cox proportional hazard regression model was utilized; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.05 to 1.81] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Pharmacokinetics of Inotuzumab Ozogamicin in Combination With Rituximab
Time Frame: 0, 1, 168 hours on Cycle 1, 2; 0, 1, 2, 168 hours on Cycle 3, 4
Population: Data for this outcome measurement was not collected since pharmacokinetic parameters were not analyzed in this study due to very few number of participants with PK samples.
Arm/Group | Rituximab + Inotuzumab Ozogamicin | Control Regimens R-CVP + R-FND
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in QT Interval Findings
Description: Assessments of QT interval was performed only in rituximab + inotuzumab ozogamicinin group. QT interval corrected using Fridericia's formula (QTcF) and Bazett's formula (QTcB) was analyzed as per common terminology criteria for adverse events (CTCAE) version 3.0, where Grade 1 = mild AE, Grade 2 = moderate AE, Grade 3 = severe AE, Grade 4 = life-threatening or disabling AE, Grade 5 = death related to AE. Number of participants with change in CTCAE grading at post-baseline time point compared to the baseline were presented. The post-baseline value was defined as the maximum grade after the first dose date on or before the end of treatment.
Time Frame: Baseline up to 42 days post-treatment
Population: Safety population included all participants who received at least 1 dose of a test article. Here 'N' signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Rituximab + Inotuzumab Ozogamicin
Number analyzed (Participants) | 9
participants
  QTcB: BL normal, post-BL normal | 4
  QTcB: BL normal, post-BL Grade 1 | 2
  QTcB: BL normal, post-BL Grade 2 | 3
  QTcF: BL normal, post-BL normal | 6
  QTcF: BL normal, post-BL Grade 1 | 3

6. Other Pre Specified Outcome: Number of Participants With Grade 3 or 4 Treatment Emergent Adverse Events (TEAEs)
Description: AE=any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Grade 3 (Severe) events=unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment. Grade 4 (Life-threatening) events caused participant to be in imminent danger of death. TEAE=between first dose of study drug and up to 42 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 42 days post-treatment
Population: Safety population included all participants who received at least 1 dose of a test article (either rituximab + inotuzumab ozogamicin or control regimens R-CVP + R-FND).
Measure: Number; unit: participants
Arm/Group | Rituximab + Inotuzumab Ozogamicin | Control Regimens R-CVP + R-FND
Number analyzed (Participants) | 15 | 13
participants | 12 | 13

7. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Findings
Description: Criteria for laboratory test abnormality: Blood Chemistry (alkaline phosphatase [greater than{>}5*upper limit of normal {ULN}, calcium [less than {<}1.75 millimole per liter {mmol/L}, creatinine [>3*ULN], glucose [>13.9 mmol/L], phosphorous [<0.6 mmol/L], potassium [<3 mmol/L], aspartate transaminase [>5.0*ULN], total bilirubin [>3*ULN]), Coagulation (international normalized ratio [>2*ULN]), Hematology (hemoglobin [<80 grams/Liter], lymphocytes [<0.5*10^9/L], absolute neutrophil count [<1*10^9/L], platelet count [<50*10^9/L], WBC [<2.0*10^9/L]).
Time Frame: Baseline up to 42 days post-treatment, disease follow up (every 12 weeks for a minimum of 1 year and up to 2 years)
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Rituximab + Inotuzumab Ozogamicin | Control Regimens R-CVP + R-FND
Number analyzed (Participants) | 15 | 13
participants
  Baseline up to 42 days post-treatment | 11 | 12
  Disease follow up | 8 | 7

8. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Criteria for determining significant change from baseline in vital signs abnormalities: heart rate value of <40 beats per minute and value >150 beats per minute, systolic blood pressure (SBP) of <80 or >210 millimeter of mercury (mmHg), diastolic blood pressure (DBP) of <40 or >130 mmHg, temperature <32 or >40 degree centigrade, and body weight>=10% increase or decrease of body weight in kilogram (kg).
Time Frame: Baseline up to 42 days post-treatment, disease follow up (every 12 weeks for a minimum of 1 year and up to 2 years)
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Rituximab + Inotuzumab Ozogamicin | Control Regimens R-CVP + R-FND
Number analyzed (Participants) | 15 | 13
participants
  Baseline up to 42 days post-treatment | 0 | 1
  Disease follow up | 3 | 2

ADVERSE EVENTS:
Time Frame: Baseline up to 42 days post--treatment
Description: Same event may appear as both AE and SAE, the presented events are distinct.Event may be serious in 1 subject and nonserious in another,or 1 subject may have experienced both SAE and non-SAE during study.TEAE=from first study drug dose up to 42 days after last dose,were absent before treatment or that worsened relative to pretreatment state.
Arm/Group | Rituximab + Inotuzumab Ozogamicin | Control Regimens R-CVP + R-FND
Serious Adverse Events (participants affected / at risk) | 6/15 | 6/13
Other Adverse Events (participants affected / at risk) | 15/15 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Inotuzumab Ozogamicin (N=15) | Control Regimens R-CVP + R-FND (N=13)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Venoocclusive liver disease (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Pneumonia cryptococcal (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Inotuzumab Ozogamicin (N=15) | Control Regimens R-CVP + R-FND (N=13)
Anaemia (Blood and lymphatic system disorders) | 2 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 5
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 2
Monocytosis (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 7
Atrial fibrillation (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 2 | 1
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1
Eye disorder (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 7
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Asthenia (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 3 | 0
Fatigue (General disorders) | 6 | 3
Feeling cold (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Pain (General disorders) | 1 | 2
Pyrexia (General disorders) | 6 | 3
Thirst (General disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 3
Bronchitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 2
Localised infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 4 | 2
Aspartate aminotransferase increased (Investigations) | 6 | 2
Bilirubin conjugated increased (Investigations) | 1 | 0
Blood albumin decreased (Investigations) | 2 | 2
Blood albumin increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 5 | 2
Blood amylase increased (Investigations) | 1 | 0
Blood bicarbonate decreased (Investigations) | 1 | 0
Blood bicarbonate increased (Investigations) | 1 | 0
Blood calcium decreased (Investigations) | 1 | 2
Blood chloride decreased (Investigations) | 1 | 0
Blood chloride increased (Investigations) | 1 | 0
Blood creatinine decreased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 3
Blood lactate dehydrogenase decreased (Investigations) | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 3 | 1
Blood phosphorus decreased (Investigations) | 0 | 1
Blood phosphorus increased (Investigations) | 2 | 3
Blood potassium decreased (Investigations) | 0 | 3
Blood sodium decreased (Investigations) | 1 | 2
Blood sodium increased (Investigations) | 1 | 0
Blood urea decreased (Investigations) | 2 | 0
Blood urea increased (Investigations) | 2 | 2
Blood uric acid decreased (Investigations) | 1 | 0
Blood uric acid increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 0
Haemoglobin decreased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
PCO2 decreased (Investigations) | 1 | 0
PCO2 increased (Investigations) | 1 | 0
Protein total decreased (Investigations) | 2 | 1
Red blood cell count decreased (Investigations) | 1 | 0
Urine output decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1
Hypouricaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 6 | 2
Memory impairment (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 3
Chromaturia (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Study did not met estimated enrollment of approximately 978 participants,thus analysis and conclusions were limited by small number of enrolled participants.Termination was not prompted by identification of safety concerns with inotuzumab ozogamicin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.